CLINICAL TRIAL: NCT00308620
Title: A Randomized, Pilot Study of the Anti-Viral and Anti-Inflammatory Effects of Chloroquine in Early HIV Infection
Brief Title: Investigating the Anti-Human Immunodeficiency Virus (HIV) & Anti-inflammatory Effect of Chloroquine
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Insufficient financial support; lack of efficacy for primary endpoint
Sponsor: University of Minnesota (Other)
Collaborators: Minnesota Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0510M77007
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: HIV Infections
Keywords: HIV; chloroquine; disease progression; inflammation; treatment naive
MeSH Terms: conditions — HIV Infections; Disease Progression; Inflammation | interventions — chloroquine diphosphate; Chloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine (Experimental): Chloroquine 205mg or 500mg orally once daily (Results pooled)
  Interventions: Drug: chloroquine phosphate
- Placebo (Placebo Comparator): Placebo once daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: chloroquine phosphate — 250mg or 500mg PO (by mouth) QDay
  Other Names: Aralen
  Arms: Chloroquine
Drug: Placebo — Placebo once daily for 8 weeks
  Arms: Placebo

SUMMARY:
Summary: Chloroquine is a medication that in laboratory settings has significant anti-HIV effects in HIV infected T-cells. Chloroquine has been used safely for over 60 years for malaria treatment and prevention, and it also has significant anti-inflammatory effects. No formal study of chloroquine has been performed in people with HIV infection. Chloroquine is used worldwide and is quite inexpensive outside of the United States. If shown to be effective, chloroquine could be a very important tool worldwide in delaying HIV disease progression which would extend the time period without needing anti-retroviral therapy. In countries where anti-retroviral therapy is not available, this could be very helpful.

This is an 8 week trial study requiring 3 study visits. Participants will be ask to take a once a day study medication (chloroquine or placebo) for 8 weeks and have three blood draws for CD4 counts, HIV viral loads, and other research tests. The visits are at study enrollment, 4 weeks, and 8 weeks.

DETAILED DESCRIPTION:
Summary:

A phase I randomized, double-blind, placebo controlled trial to investigate the efficacy of chloroquine to decrease T-cell activation and decrease viral load in early HIV.

Scientific Rationale:

Chloroquine has in vivo direct anti-HIV effects and an anti-inflammatory effect. These properties may be beneficial in reducing viral burden and immune activation therefore delaying HIV disease progression.

Sample Size: 25

Length of Study: 8 weeks, [enrollment + 2 follow up visits].

Intervention:

* Arm 1a: Chloroquine 250mg orally once daily for 8 weeks.
* Arm 1b: Chloroquine 500mg orally once daily for 8 weeks.
* Arm 2: Placebo once daily for 8 weeks.

Measurements:

* Blood draws at weeks: 0, 4, and 8 weeks.
* CD4, viral load measurements will be communicated to the referring provider (with subject consent).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults
* CD4 count > 250 cells/mm3
* Not presently receiving HIV antiretroviral therapy (> 6 months or naïve)
* Viral load > 3000 RNA copies/mL (3.5 log)
* No planned HIV anti-retroviral therapy for 8 weeks

Exclusion Criteria:

* Prior retinal eye disease
* CD4 < 250 cells/µL
* Renal failure
* Active malignancy
* Corticosteroid therapy
* Age < 18 or > 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Boulware, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- Minnesota ACTU, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Murray SM, Down CM, Boulware DR, Stauffer WM, Cavert WP, Schacker TW, Brenchley JM, Douek DC. Reduction of immune activation with chloroquine therapy during chronic HIV infection. J Virol. 2010 Nov;84(22):12082-6. doi: 10.1128/JVI.01466-10. Epub 2010 Sep 15. PMID 20844049
- See also: University of Minnesota Clinical Virology Program — http://cvp.umn.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2006-2008 recruitment of volunteers in HIV care but electing to not receive ART.
Groups:
- Chloroquine 500mg: Chloroquine 500mg PO once daily x 8 weeks
- Chloroquine 250mg: Chloroquine 250mg PO once daily x 8 weeks
Period: Overall Study
Arm/Group | Chloroquine 500mg | Placebo | Chloroquine 250mg
Started | 3 | 4 | 6
Completed | 2 | 3 | 5
Not Completed | 1 | 1 | 1
Not completed — Death | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroquine 500mg | Placebo | Chloroquine 250mg | Total
Number analyzed (Participants) | 3 | 4 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 6 | 13
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (15) | 34 (5) | 36 (5) | 36.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 3 | 3 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: HIV Viral Load Change
Description: HIV-1 viral load change between baseline and 8 weeks
Time Frame: baseline and 8 weeks
Measure: Log Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Chloroquine 250mg or 500mg: Chloroquine 250mg or 500mg orally once daily x 8 weeks. n=6 for 250mg; n=3 for 500mg
- Placebo: Placebo orally once daily for 8 weeks
Arm/Group | Chloroquine 250mg or 500mg | Placebo
Number analyzed (Participants) | 9 | 4
log10 copies/mL | -.083 (.5) | 0.0 (.1)

2. Secondary Outcome: Change in Immune Activation Assessed by Flow Cytometry Analysis From Baseline to 8 Weeks
Description: The Change in the percentages of CD38+ HLA-DR+ CD8 and CD4 memory T cells from baseline to 8 weeks.
Time Frame: 8 weeks
Population: Analysis of Chloroquine arms is pooled.
Measure: Median (Full Range); unit: percentage change
Groups:
- Chloroquine 250mg or 500mg: Chloroquine 500mg orally once daily x 8 weeks
Arm/Group | Chloroquine 250mg or 500mg | Placebo
Number analyzed (Participants) | 7 | 3
percentage change
  CD8 CD38+HLA-DR+ | -2.5 [-7 to 2] | 1.85 [-3 to 2]
  CD4 ki67+ | -2.0 [-3 to 2] | 1.4 [-0.5 to 3]

ADVERSE EVENTS:
Arm/Group | Chloroquine 500mg | Placebo | Chloroquine 250mg
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroquine 500mg (N=3) | Placebo (N=4) | Chloroquine 250mg (N=6)
Death (non-related) (Social circumstances) | 1 (1) | 1 (1) | 0 (0) — Autopsy Report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No